CLINICAL TRIAL: NCT04857008
Title: Phase II Pilot Study Evaluating the Feasibility of Delivery and Evaluation of BNT001, a Digital Cognitive-Behavioral Stress Management (CBSM) Software Application for Treatment of Anxiety and Depressive Symptoms in Veterans With Cancer
Brief Title: BNT001 Digital Therapeutic Feasibility Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment challenges
Sponsor: Blue Note Therapeutics (Industry)
Collaborators: Durham VA Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: BNT001 VA Pilot Study_3_4_2021
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BNT001 (Experimental): BNT001 is a commercially-available, prescription-only, software / medical device in the form of a digital application (digital app) for use on the participant's mobile device which delivers 10-sessions on cognitive behavioral therapy for cancer patients.
  Interventions: Device: BNT001

INTERVENTIONS:
Device: BNT001 — BNT001 is a commercially-available, prescription-only, software / medical device in the form of a digital application (digital app) for use on the participant's mobile device which delivers 10-sessions on cognitive behavioral therapy for cancer patients.

SUMMARY:
This single arm phase II trial focused on cancer patients and cancer survivors in the Veterans Health Administration will gather data on feasibility, acceptability, ease of clinical implementation, and preliminary efficacy of BNT001, a prescription digital software application. BNT001 delivers a 10-session digitally administered version of a published manualized therapy for stress management in adult cancer patients that has established efficacy in improving quality of life and mood.

DETAILED DESCRIPTION:
This pilot will study specific implementation barriers and facilitators, procedures that are necessary to ensure adherence to utilization of the digital program, as well as any potential safety issues associated with recruiting and offering an intervention to cancer patients with moderate anxiety or mild depressive symptoms. Data relating to patient experience, adherence, satisfaction and pre-post intervention outcomes will also be tracked.

The study will run in two distinct phases to first assess the process of clinical implementation by prescribing oncology clinicians, and in a second more expanded phase, further assess the clinical implementation and impact on enrolled patients.

Study Phase 1: We aim to identify promoters and barriers to the clinical implementation of BNT001, a software application that delivers a 10-session digitally administered version of a published manualized therapy for stress management in adult cancer patients that has established efficacy in improving quality of life and mood.

Study Phase 2: We aim to further identify promoters and barriers to provider clinical implementation of BNT001, assess patient acceptability and feasibility including patient adherence to BNT's 10-sessions, and obtain preliminary data on BNT001's impact on cancer-related distress.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis or history of invasive cancer (excluding non-melanoma skin cancer).
* Patients showing mild to moderate anxiety or depression on the Veteran System Assessment Screen (VSAS), with anxiety or depression scored as 1-6 on a 0-10 scale.
* Fluent in English.
* Has access to iOS or Android smartphone, or tablet and capable of receiving text messages.
* Has an e-mail address.

Exclusion Criteria:

* Endorses thoughts of self-harm, history of suicidality.
* Currently participating in investigative behavioral intervention trial for treatment of anxiety or depression.
* Participant is unable to complete training, has cognitive deficits, major psychiatric conditions, psycho-social conditions; lack of access to reliable internet and accessible device; other social conditions that would interfere with adherence to self directed care, such that in investigator's opinion the participant would be unable to complete the study.
* Recently completed use of Blue Note Therapeutics COVID Cancer Care Program or other Blue Note Therapeutics sponsored study.

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Identification of promoters and barriers to clinical implementation | Baseline to 4 weeks
  Identification of promoters and barriers to clinical implementation of BNT001, a software application that delivers a 10-session, cancer-specific, behavioral intervention called Cognitive-Behavioral Stress Management (CBSM), to adult patients currently undergoing cancer treatment.
To measure changes in pre and post cancer-related distress in patient participants. | Baseline to 12 weeks
  Patient participants symptoms will be assessed with the Veterans Symptom Assessment Screen (VSAS). The VSAS is a clinical patient reported outcomes tool to document cancer-related symptoms to improve quality of life that has been adopted across VA hematology-oncology sites. The VSAS is comprised of 13 symptoms, rated on a 0 to 10 scale.

SECONDARY OUTCOMES:
Patient completion rates | Baseline to 12 weeks
  To measure patient completion rates via the BNT001's underlying device data capture system.
Patient feasibility and acceptability | Baseline to 12 weeks
  To measure patient feasibility and acceptability via a midpoint and post-completion questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Friedman, MD, Principal Investigator — Durham Veterans Administration Health Care System
Locations (1):
- Durham Veterans Administration, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No